CLINICAL TRIAL: NCT02451384
Title: To Compare the Influences of Different Methods to Remove the Pancreatic Ductal Adenocarcinoma With the Detection of Circulating Tumor Cells
Brief Title: According CTC to Compare the Influences of Different Methods to Remove the PDAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Wenhui Lou, Associate Professor of General Surgery Department, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2015-010
Record Dates: First submitted 2015-05-14; First posted 2015-05-22 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-06

CONDITIONS: Carcinoma, Pancreatic Ductal; Circulating Tumor Cells
MeSH Terms: conditions — Carcinoma, Pancreatic Ductal; Neoplastic Cells, Circulating | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- routine surgery (Experimental): In this arm the patients will be performed routine surgery to remove the tumors. And then we compare their circulating tumor cell countings in the pre and post-operation.
  Interventions: Procedure: routine surgery
- no-touch surgery (Experimental): In this arm the patients will be performed no-touch surgery to remove the tumors. And then we compare their circulating tumor cells countings in the pre and post-operation.
  Interventions: Procedure: no-touch surgery
- laparoscopy surgery (Experimental): In this arm the patients will be performed laparoscopy surgery to remove the tumors. And then we compare their circulating tumor cells countings in the pre and post-operation.
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: routine surgery — To observe if the surgeries can influence the countings of circulating tumor cells of the patients.
  Arms: routine surgery
Procedure: no-touch surgery
  Arms: no-touch surgery
Procedure: laparoscopic surgery
  Arms: laparoscopy surgery

SUMMARY:
Acccording circulating tumor cells to compare the differences of different methods(routine method、no-touch principle method、laparoscopy method) to remove the ductal adenocarcinoma of pancreatic body and tail.

ELIGIBILITY:
Inclusion Criteria:

* Ductal adenocarcinoma of pancreatic body and tail
* Tumor can be removed
* No other tumors and without liver metastases
* Age from 18 to 80 years old

Exclusion Criteria:

* Neoplasms with other sites of the pancreas
* With other tumors of any other sites

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the changes of CTCs countings between the pre and post-operation in each arm | Within 1 week after the surgeries are completed in any arm
the changes of CTCs countings between the pre and post-operation among the arms | Within 2 weeks after the surgeies are all completed

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Genaral surgery department of Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality